CLINICAL TRIAL: NCT02102737
Title: Comparaison d'Une Nouvelle Technique de Mesure de l'insulinorésistance Par Scintigraphie Avec la Technique de référence : Utilisation du 6-DIG Comme Marqueur du Transport du Glucose.
Brief Title: Comparison of A New Technique of Measure of the Insulin Resistance By Scintigraphy With the Reference Technique
Acronym: GLUCIMAG2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C13-14; 2013-003526-92 (EudraCT Number)
Record Dates: First submitted 2014-03-25; First posted 2014-04-03 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus; Insulin Resistance; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases
Keywords: insulin resistance; Scintigraphy; Hyperinsulinemic euglycemic clamp
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — Constriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 6-DIG and clamp (Experimental): injection of 6-DIG and hyperinsulinemic euglycemic clamp
  Interventions: Drug: 6-DIG; Procedure: clamp

INTERVENTIONS:
Drug: 6-DIG — injection of 6-DIG
Procedure: clamp — hyperinsulinemic euglycemic clamp

SUMMARY:
Insulin resistance is closely associated with apparition of type 2 diabetes mellitus; it is an independent risk factor and predicts future cardiovascular events.

Hyperinsulinemic euglycemic clamp is a validated method to assessment of insulin resistance and It is also the gold standard technique. However, the complexity and length of this technique render it unsuitable for routine clinical use.

In this study, the investigators use a new technique to provide precise, objective, fast and automated quantification of insulin resistance with camera SPECT.

They compare the results with those of the measurement of hyperinsulinemic euglycemic clamp in population with or without insulin resistance.

The proposed study is to validate this new non-invasive imaging technique for evaluation of insulin resistance in patients with or without insulin resistance with a comparison with hyperinsulinemic euglycemic clamp.

DETAILED DESCRIPTION:
Currently, type II diabetes mellitus, has reached epidemic levels in the world. Moreover, the prediction for the year 2030 is even more alarming. Insulin resistance, characterized by a depressed cellular sensitivity to insulin in insulin-sensitive organs, is a central feature of the metabolic syndrome and a risk factor for type 2 diabetes. Its appearance may precede the diagnosis of true diabetes several years. Insulin resistance results in decreased membrane translocation of GLUT-4, whole the molecular mechanism remains unclear. Currently, there is no simple tool to measure insulin resistance. The gold standard technique remains the hyperinsulinemic euglycemic clamp. However, the complexity and length of this technique render it unsuitable for routine clinical use. Many methods or index have been proposed to assess insulin resistance in human, but none have shown enough relevance to be used in clinical use. Moreover, all these clinical measurements focus on whole-body glucose uptake, however an accurate and convenient procedure for insulin resistance measurement by organ would be interesting. Indeed there are increasingly evidences to insulin resistance as a primary etiologic factor in the development of nonischemic heart failure (HF), another growing public health problem.

Nuclear imaging provides interesting methods to measure insulin resistance using Positron Emission Tomographic (PET) tracer. Two glucose analogs [18F]2-fluoro-2-deoxy-D-glucose (FDG) and [11Cl-30methyl-n-glucose (3-OMG) have been used to evaluate noninvasively the cellular uptake of glucose using PET techniques for several organs like heart, skeletal muscle blood-brain barrier, and liver. [18F] 2-fluoro-2-deoxy-D-glucose (FDG), the most commonly used to study glucose metabolism in humans, allows the estimation of glucose transport and its phosphorylation. A number of kinetic modeling approaches have been used for the quantitation of glucose utilization rates using FDG. FDG is transported and phosphorylated as native glucose, but calculation of glucose uptake and metabolism requires the use of correction factors for each process merged into a lumped constant. The major limitation of these approaches is that quantification of glucose metabolism requires the knowledge of the lumped constant, a factor, which relates the kinetic behavior of FDG to naturally occurring glucose in terms of the relative affinity of each molecule for the trans-sarcolemmal transporter and for hexokinase. Unfortunately, the value of the lumped constant in humans under different physiological and pathophysiological conditions varies, and metabolic imaging with PET need standardization of metabolic conditions by hyperinsulinaemic euglycaemic clamp. 3-OMG appears as an ideal glucose analog to probe transmembrane transport. However, due to the short half-life of the 11C (t1/2 = 20 min), this analog can be used only in clinical institutions in close proximity of a cyclotron and which have access to PET devices.

According to these knowledge, the investigators have developed an original compound, [123I] 6-deoxy-6-iodo-D-glucose (6DIG), as a tracer of glucose transport equivalent to 3-OMG, the reference tracer. 6-DIG has previously been exploited to measure IR in vivo and the investigators transfer to human this measurement technique, perfectly validated in animal. Previous, they have reported the first use a potential single-photon emission computed tomography (SPECT) tracer to study basal and insulin-stimulated glucose transport non-invasively. In a phase I of development, they use a new nuclear probe using an iodinated tracer of glucose transport for clinical application and specific imaging processing to assess cardiac insulinoresistance in healthy or diabetic subjects. The results in human subjects show that this technique rapidly provides insulinoresistance index (ratio scintigraphy measurement of glucose transport in heart before and after infusion of insulin) in a simple procedure, opening up new opportunities for screening for pre-diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Insulin sensible patients

  * Body mass index < 25 HOMA <= 2.5
  * Waist measurement < 94 cm for men and < 80 cm for women
  * HDL cholesterol 1,03 mmol/L for men and > 1,29 mmol/L for women
  * Triglyceride level ≤ 1,69 mmol/ L
  * For women not menopausal since at last one year or not surgically sterilised:

On-going contraception, physical or hormonal, excepted local methods (spermicidal, diaphragm, condom, cape)

- Insulin resistant patients

* For women not menopausal since at last one year or not surgically sterilised:
* On-going contraception, physical or hormonal, excepted local methods (spermicidal, diaphragm, condom, cape)
* HOMA > 2.5
* Body mass index > 25
* Waist measurement > 94 cm for men and > 80 cm for women
* HDL cholesterol < 1,03 mmol/L et for men and ≤ 1,29 mmol/L for women
* Triglyceride level > 1,69 mmol/ L

Exclusion Criteria:

* • Instable cardiomyopathy

  * Severe hypertension defined by par SAP > 180 mmHg and/or DAP > 110 mmHg
  * Psychiatric illness, needing a chronic treatment
  * Previous history of stroke, epilepsy, cranial trauma, pituitary surgery, disease likely to reduce the ability of absorption, diffusion or excretion of the radiotracer.
  * Allergy to one of the components of the products used during the study
  * Treatment likely to interfere with glucose metabolism
  * Alcohol or drug intoxication
  * Vegetarian or restrictive low-calory diet,
  * Participation in other biomedical research at the same time or exclusion period under another biomedical research
  * Pregnant, parturient or breast-feeding women,
  * Inappropriate way of life

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05-13 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Correlation between measure of insulin resistance measurement by scintigraphy and hyperinsulinemic euglycemic clamp | DAY 1 AND DAY 2
  Correlation between measure of insulin resistance measurement by scintigraphy (insulin resistance index: ratio scintigraphy measurement of glucose transport in heart before and after infusion of insulin) and hyperinsulinemic euglycemic clamp (Glucose Infusion Rate and sensibility index Clamp)

SECONDARY OUTCOMES:
SAFETY | visit 2, visit 3 and visit 4
  A systematic collection of adverse events
Reproducibility | day 2 and day 3
  Reproducibility inter and intra operator of Insulin resistance index
Left ventricule ejection fraction | day 2
left ventricle volume | day 2
cardiac mass | day 2
diastolic function | day 2
cardiac output | day 2
pulmonary pressure and right ventricular function | day 2
strain by speckle tracking echocardiography | day 2

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Barone-Rochette, PHU, Principal Investigator — Hopital Michalon , CHU de Grenoble
Locations (1):
- Hôpital Michallon . CHU Grenoble, Grenoble, France